CLINICAL TRIAL: NCT03302390
Title: Role of Chemokine and Chemokine Receptor in Psoriasis
Status: Withdrawn | Type: Observational
Why Stopped: PI failed to submit study for continuing review by IRB
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1015909; 5R01AR063091 (NIH)
Record Dates: First submitted 2017-07-08; First posted 2017-10-05 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Biopsy; Injections; Lidocaine; Epinephrine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biopsy of Skin with Psoriasis: Shave biopsy of psoriasis lesion
  Interventions: Procedure: Shave Biopsy of Psoriasis Lesion

INTERVENTIONS:
Procedure: Shave Biopsy of Psoriasis Lesion — The investigator will take about 0.5x0.5 inch square section of skin from the psoriasis lesion. To numb the skin, the subject will receive a small injection of 0.5% lidocaine HCl 5mg/mL with 1:200,000 mcg/mL epinephrine solution as per standard shave biopsy protocol. The shaving instrument has a blade that will shave off a superficial piece of skin that is less than <3mm in thickness. After 14 days, the subject will return to make sure that the skin biopsy site has healed properly. The piece of skin that is removed will be grafted onto the back of an immunocompromised SCID mouse. An approved IACUC protocol covering this procedure will be in place prior to engraftment.
  Other Names: shave biopsy; biopsy; injection, lidocaine HCl with epinephrine

SUMMARY:
This study aims to elucidate the role of Chemokine and chemokine receptor in the pathogenesis of Psoriasis by using human psoriasis skin xenograft SCID mouse model. The hypothesis is that chemokine and chemokine receptor play important roles in psoriasis and establishment of human skin xenograft mouse model provide excellent platform to test the hypothesis.

DETAILED DESCRIPTION:
Chemokines belongs to a large group of small chemotactic proteins (8-11 kilodaltons in size). Upon engagement of chemokine, chemokine receptor can activate downstream intracellular signaling pathways and results in diverse cellular processing such as cytoskeleton reorganization and cell locomotion. Chemokines are chemoattractant factors and can stimulate directional migration of all classes of leukocytes such as T cells. Epidermal keratinocytes in the skin are able to express multiple chemokines that can attract certain leukocytes, such as T cells or dendritic cells (DCs), to migrate to the epidermis. Psoriasis is a type of skin inflammatory diseases that results in misregulated immune system including immune cell infiltration. Keratinocyte secreted chemokine and chemokine receptor on leukocytes have been known to involve in the pathogenesis of psoriasis. However, it is not very clear how chemokines are regulated in keratinocytes and the binding of chemokine to receptor on leukocytes controls the pathogenesis of psoriasis. To better understand the immune regulation of chemokine and chemokine receptor in the molecular mechanism and pathogenesis of psoriasis, the investigators plan to establish human psoriasis skin xenograft mouse model that involves graft of human skin onto immune deficient mice. The human skin, including lesional and non-lesional skins, has been proven to be acceptable to the SCID mice and the phenotype can maintain for a number of months. The advantage of the xenograft model is to that it can preserve the full complexity of human diseases and thus resembles the pathogenesis of human diseases. This model has also been shown with constant efficacy of anti-psoriasis drug in comparison with clinical practice. Thus, this mouse model has great value to help the investigators understand how chemokine and immune cells are regulated in psoriasis. Of particular note is that this model can be used to test therapeutic drug before introduce them into clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or greater
* Subjects need to fulfill the diagnostic evidence of psoriasis with or without psoriatic arthritis
* Subject may take the following medicines: NSAID, hydroxychloroquine, sulfasalazine, prednisone (<10 mg/day), Methotrexate (10 mg/week)
* Subject needs to stop topical skin preparations other than emollients in one small plaque of psoriasis for 3-4 wks from where the shave biopsy will be taken
* Willing and able to provide informed consent in English

Exclusion Criteria:

* Subjects less than 18 years old
* no clinical evidence of psoriatic skin
* Subjects with contraindications for biopsy, and patients receiving anticoagulants
* Subjects with active hepatitis B or Hepatitis C infection
* Subjects with concomitant inflammatory diseases such as inflammatory bowel disease, gout
* Subjects who are taking the following systemic biological therapies for psoriasis: cyclosporine, methotrexate, prednisone, acitretin, sulfasalazine, certolizumab, etanercept, adalimumab, infliximab, golimumab, secukinumab, ustekinumab, and apremilast. Other systemic medications may exclude the subject from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or greater will be recruited for this study. The study population will include patients at UC Davis Dermatology with diagnostic evidence for psoriasis who do not have coexisting inflammatory diseases.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Acquisition of psoriatic skin from patient to transfer to immunocompromised mice | Five years
  The purpose of this human clinical trial is to harvest psoriatic skin for engraftment onto immunocompromised mice. The primary outcome measure is to identify a 0.75 x 0.75 square inch piece of skin with psoriasis on study subjects to be biopsied. specific outcome measure that will be obtained in the patients other than ensuring that their graft sites heal appropriately. Their skin, once placed on immunocompromised mice, will be used to test new therapeutic drugs which might have a beneficial outcome in psoriasis, as measured in this mouse model.

SECONDARY OUTCOMES:
Observe Appropriate Healing in Subject Biopsy sites | Five years
  The secondary outcome measure is to observe that study subjects' graft sites heal appropriately.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Hwang, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No